CLINICAL TRIAL: NCT02404766
Title: Effects of C0-C1 Mobilization in the Neutral Position in Subjects With Upper Cervical Rotational Hypomobility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, César Hidalgo, Unidad de Investigación en Fisioterapia, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP23/2012
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Upper Cervical Spine Rotational Hypomobility
Keywords: manual therapy; cervical; range of movement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Intervention group (Experimental): C0-C1 dorsal glide mobilization in the cervical neutral position.
  Interventions: Other: C0-C1 dorsal glide manual mobilization
- Intervention group 2 (Experimental): C7-T1 ventral cranial glide mobilization in the cervical neutral position
  Interventions: Other: C7-T1 ventral cranial glide manual mobilization
- Control group (No Intervention): Not receiving any intervention

INTERVENTIONS:
Other: C0-C1 dorsal glide manual mobilization
  Arms: Intervention group
Other: C7-T1 ventral cranial glide manual mobilization
  Arms: Intervention group 2

SUMMARY:
C1-C2 is the most mobile segment of the spine and its dysfunction is frequently associated to cervical pain and headache. However, serious neurovascular adverse effects have been documented through direct treatment of C1-C2 segment. Although indirect treatment via adjacent segments and avoidance of end range of rotation and extension have been recommended for a safer and effective cervical treatment, there is no scientific evidence of the effectiveness of the indirect treatment approach in the cervical neutral position for C1-C2 hypomobility.

Due to that, the investigators designed a randomized controlled trial to compare the short-term effects in the Flexion Rotation Test (FRT) of a translatoric mobilization of C0-C1, a translatoric mobilization of C7-T1 and a control group in subjects with C1-C2 hypomobility.The primary hypothesis is that C0-C1 dorsal glide mobilization applied in the neutral cervical position can recover the C1-C2 rotational range of movement in subjects with upper cervical hypomobility.

ELIGIBILITY:
Inclusion Criteria:

* FRT with less than 32º or asymmetry of 10º between right and left, whenever one of the sides does not exceed physiological C1-C2 ROM (45º)
* Indication of grade III mobilization in C0-C1 and C7-T1 segments
* Aged 18-66
* Signed informed consent

Exclusion Criteria:

* Contraindication to manual therapy and red flags according to Rushton et al. (2012)
* Pain presence at the beginning or during the study
* Cervical treatment during the last three months
* Inability to tolerate FRT
* Involvement in litigation or compensation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in baseline in Range of movement in Upper Cervical Spine | 1 hour after intervention
  Flexion-rotation test measured by CROM device

SECONDARY OUTCOMES:
Cervical range of movement in cardinal planes | 1 hour after intervention
  Active cervical range of movement in sagittal, frontal and transversal planes measured by CROM device.
Upper cervical flexion and extension range of movement | 1 hour after intervention
  Active upper cervical flexion and extension range of movement measured with CROM device

CONTACTS AND LOCATIONS:
Locations (1):
- César Hidalgo, Zaragoza, Aragon, Spain